CLINICAL TRIAL: NCT00932178
Title: Calmer Life: A Worry Reduction Program for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Melinda Stanley, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRECC006; VA ID Number: 09E02.H (Other: MEDVAMC Research & Development Committe)
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Anxiety
Keywords: Anxiety; Worry; nervousness; Older Adult
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calmer Life (Experimental): Skills-based intervention to reduce anxiety and worry in adults age 50+.
  Interventions: Behavioral: Calmer Life

INTERVENTIONS:
Behavioral: Calmer Life — Calmer Life is a modified version of an existing Cognitive Behavioral Treatment manual. Participants have the option of including religion and spirituality into coping skills taught as a way of treating anxiety with or without depression in older adults.

SUMMARY:
Calmer Life is a research study for older adults with anxiety. In the program participants will have the opportunity to learn skills that may help cope with anxiety. Participants have the option of including religion and spirituality into the skill. Skills participants can learn include: how to relax, how to change the way you think about things, and how to solve problems more effectively.

DETAILED DESCRIPTION:
Preliminary work in a related study (H-22763) suggests that a significant percentage of older patients think that incorporating religion and/or spirituality into counseling is important. Based on data from this study, available scholarly literature, and input from consultants, we have developed an initial version of Calmer Life that is sufficiently flexible to incorporate a range of religious and spiritual beliefs and coping skills based on each patient's unique values and beliefs. The manual for this treatment includes intervention components from evidence-based treatment for late-life anxiety (H-23798; H-15958), suggested strategies for incorporating religion or spirituality into the coping skills for anxiety and depression, and spiritually-based interventions (e.g., forgiveness, gratitude). Patients have a choice to include or not include religious or spiritually based components. The proposed project will begin to test this broad spiritually based CBT for older adults (Calmer Life) with Generalized Anxiety Disorder (GAD) with or without depression. Further modifications to the Calmer Life manual and in the treatment approach will be made based on patient, clinician, and consultant input.

ELIGIBILITY:
Inclusion Criteria:

* Age 50+;
* A principal or co-principal diagnosis of General Anxiety Disorder;
* Interest in receiving CBT for anxiety/depression with the option of including religion and spirituality;
* Must be English speaking

Exclusion Criteria:

* Active suicidal intent;
* Current psychosis or bipolar disorder;
* Substance abuse within the last month

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Geriatric Depression Scale (GDS), Geriatric Anxiety Inventory (GAI), Penn State Worry Questionnaire (PSWQ-A), State-Trait Anxiety Inventory (STAI) | Baseline, 1-month, 2-month, 3-month, and 6-month

CONTACTS AND LOCATIONS:
Overall Officials: Melinda A. Stanley, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E DeBakey VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Background] Jameson JP, Shrestha S, Escamilla M, Clark S, Wilson N, Kunik M, Zeno D, Harris TB, Peters A, Varner IL, Scantlebury C, Scott-Gurnell K, Stanley M. Establishing community partnerships to support late-life anxiety research: lessons learned from the Calmer Life project. Aging Ment Health. 2012;16(7):874-83. doi: 10.1080/13607863.2012.660621. Epub 2012 Mar 15. PMID 22416908